CLINICAL TRIAL: NCT05659394
Title: Intermittent Pneumatic Compression of the Thigh for the Treatment of Lower Limb Wounds: a Randomised Control Trial
Brief Title: Intermittent Pneumatic Compression of the Thigh
Acronym: IPCOTT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Huntleigh Healthcare Ltd (Industry)
Collaborators: SerenaGroup, Inc. (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1341779
Record Dates: First submitted 2022-12-05; First posted 2022-12-21 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Venous Leg Ulcer
MeSH Terms: conditions — Varicose Ulcer

STUDY DESIGN:
Intervention Model Description: The IPCOTT study is a parallel global multicentre, pragmatic, open, randomised controlled trial of IPC (2hrs daily) plus standard wound care vs. standard wound care alone.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Standard Wound Care Alone (Other): Patients receiving gold standard compression therapy for venous or mixed etiology ulcers
  Interventions: Other: Standard Wound Care Alone
- Standard Wound Care plus IPC (Other): Patients receiving gold standard compression therapy plus IPC (WoundExpress)
  Interventions: Device: Stand Wound Care plus IPC

INTERVENTIONS:
Other: Standard Wound Care Alone — gold standard compression therapy
  Arms: Standard Wound Care Alone
Device: Stand Wound Care plus IPC — gold standard compression therapy plus IPC (WoundExpress)
  Arms: Standard Wound Care plus IPC

SUMMARY:
Study Summary

A leg ulcer is a long-lasting (chronic) sore that takes more than two weeks to heal. The majority of leg ulcers are caused either by problems with the veins in the legs; these are called 'venous leg ulcers' (VLU), or a combination of both venous and arterial disease which affects the veins and arteries in the leg; these are called 'mixed aetiology ulcers'(MLU). Venous and mixed aetiology leg ulcers are usually treated by applying a simple non-stick dressing to the ulcer with a firm compression bandage applied on top. These bandages are designed to squeeze the legs and encourage blood flow towards the heart. Before this treatment starts, a patient may undergo tests to check the flow of blood in the leg arteries is adequate. This ensures that compression bandaging can be safely applied to assist wound healing without compromising arterial blood flow.

Most venous and mixed aetiology leg ulcers heal within three to four months if they're treated by a healthcare professional trained in compression therapy for leg ulcers. However, some ulcers can be more problematic and may persist for many months or even years despite being treated with the gold standard treatment of compression bandages. We therefore need to find more ways of helping these problematic ulcers to heal.

Intermittent Pneumatic Compression (or IPC) is another way of compressing legs to try and improve the circulation. IPC consists of a sleeve or garment which is applied to the leg. The sleeve is connected to a pump which gently inflates and then deflates it to squeeze the leg in a massage like manner.

The IPCOTT study aims to find out if a new IPC device, known as the WoundExpress can help to heal leg ulcers. The WoundExpress has a sleeve that patients put around the thigh, like the one applied to the arm when people have their blood pressure taken. Users need to be either sitting with their legs raised or lying down when using the device. Pressing the 'start' button on the pump causes the sleeve to automatically inflate with air for 2 minutes, until it reaches a pressure of 60 mm/Hg (this is low compared to the pressure used when measuring blood pressure; most patients find it very gentle and comfortable). After the 2-minute inflation, the sleeve will automatically deflate for another 2 minutes, where no compression is applied to the thigh. These 4-minute inflation and deflation cycles will repeat whilst the device is in use.

People who take part in the study will be randomly allocated to Group A or Group B. Patients in Group A will continue to receive their usual wound care but will also be provided with a WoundExpress device to use for 2 hours per day for a 16-week period. Patients in Group B will continue to receive their standard wound treatment only for the 16-week study period (patients in Group B will be offered the chance to use the WoundExpress device for a 16-week period after the study has ended). All patients taking part in the study will be asked to attend their Wound Clinic for a study review once every two weeks during the study period. At these visits, a research nurse will take measurements and photographs of the ulcer(s) and participants will also be asked some questions about how they have been feeling since using the device. Patients who have been given a WoundExpress device will also be asked to keep a diary recording when they use the device and how they found it.

When the study is complete, results will be analyzed to find out if there was any difference in ulcer healing rates between Group A and Group B.

DETAILED DESCRIPTION:
Clinical Problem:

A leg ulcer is defined as the loss of skin below the knee on the leg or the foot, which takes more than two weeks to heal. Leg ulcers are the most common wound type in the community in the UK with a prevalence rate of approximately of 0.45/1000 in men and 0.56/1000 in women, increasing to 8.29/1000 in men and 8.06/1000 in women aged over 85 years old. Leg ulcers of venous origin account for approximately 70% of individuals with leg ulcers, with 10-20% being due to a combination of venous and arterial disease, often referred to as mixed leg ulcers (MLU).

Leg ulceration represents a significant source of morbidity with adverse physical, social and psychological sequalae. With appropriate treatment, some ulcers heal successfully within a few weeks, however many persist for months and even several years. The annual cost of managing patients with venous leg ulcers alone in Wales is £7,706 per patient per annum, which translates to an annual cost of over £2 billion when extrapolated to the United Kingdom (UK) population.

Current Treatment Compression therapy in the form of graduated, multi-layered bandaging, is widely accepted as the treatment of choice and gold standard therapy for the prevention and management of VLU. Compression therapy can also be recommended for mixed aetiology wounds where vascular assessment has been completed and there is no evidence of severe peripheral arterial disease (PAD) whereby compression therapy would be contraindicated. Patients with mixed etiology ulceration of the lower limb with an ankle brachial pressure index (ABPI) of >0.5 and an absolute ankle pressure >60 millimeters of mercury (mmHg) were able to receive inelastic compression up to 40 mmHg without restricting arterial perfusion. Other published guidance suggests a more conservative approach to compression with mixed disease with moderate PAD, utilizing a reduced level delivering approximately 20 - 30 millimeters of mercury compression at the ankle or the use of mild to moderate compression incorporating pressures <20 millimeters of mercury up to 40 millimeters of mercury.

However, a proportion of wounds do not progress towards healing despite receiving this gold standard treatment and furthermore some patients cannot tolerate wearing continual compression bandaging. A study showed that of 440 patients with VLUs who were in gold standard compression, 48% had not healed within 12 months. Comparable healing rates between VLU and MLU treated with reduced compression have been previously demonstrated.

Physiological Effects of IPC

Application of IPC to the limb affects underlying subcutaneous tissue, muscle and blood vessels resulting in a range of physiological effects including alterations in blood flow dynamics and the release of biochemical mediators that affect the circulatory system. The effects of IPC are documented as:

* Increasing venous blood flow: When IPC is applied to the lower limb, or part of, the application of cyclical intermittent compression causes a pulsatile flow to move proximally. This drains the blood at the compression site and increases venous flow, simulating the action of the calf muscle pump. This can also facilitate clearance within the venous valve sinuses. Venous hypertension is reduced and there is a decrease in local oedema that in turn increases capillary perfusion.
* Increasing arterial blood flow: If arterial compression is applied at sufficient pressure to occlude arterial blood flow, ischemia will occur and on release of the compression, a reactive hyperemia ensues. This reactive hyperemia also occurs at lower pressures when the veins are compressed, and several mechanisms have been suggested as to why this occurs. By increasing venous flow, there is a corresponding increase in the arterio-venous pressure gradient that in turn causes an increase in arterial blood flow. Additional hypotheses include suspension of the veno-arteriolar reflex, and a myogenic mechanism. The veno-arteriolar response to an increase in venous pressure is neurally controlled. It has been suggested that the reduced venous pressure produced by mechanical compression, suppresses the veno-arteriolar reflex; allowing arterioles to dilate, and enabling a hyperemia to ensue. The proposed myogenic mechanism is a vascular response to alterations in intravascular pressures. Arteriolar smooth muscle is believed to respond directly to the increased distension that arises as a result of raised intravascular pressure by constricting; and conversely, a loss in vascular tone and hence dilation occurring in response to a decrease in intravascular pressure.
* The act of compression also increases mechanical stress on the endothelial lined wall of the artery causing a release of biochemical substances with anti-thrombotic, pro-fibrinolytic and vasodilatory properties. Hematological studies have demonstrated that patients with chronic venous insufficiency have a reduced plasma fibrinolytic activity. IPC increases tissue plasminogen activator (tPA) and urokinase-plasminogen activator (UPA) with a corresponding decrease in plasminogen activator inhibitor-1 (PAI-1). These actions have the overall effect of suppressing pro-coagulant activity whilst enhancing the fibrinolytic mechanism.

Evidence of effectiveness of IPC in the treatment of venous and mixed leg ulceration In 2014, a Cochrane review found that there was some limited evidence that showed that IPC may improve healing of venous leg ulcers when added to compression bandaging. Five trials compared IPC plus compression with compression alone. Two of these found increased healing with IPC than with compression alone. The remaining three trials (122 people) found no evidence of a benefit of IPC plus compression compared with compression alone. However, all of these trials were noted as being at high risk of bias as a result of inadequate randomization procedures, allocation concealment and blinded outcome assessments. Additional research, undertaken after this review, is limited and is confined to case report series. Another study found that IPC combined with negative pressure wound treatment appeared to promote healing and reduce associated chronic pain in 11 patients with venous leg ulcers. More recent studies have also demonstrated that IPC can improve the symptoms of arterial insufficiency and reduce oedema. Further high-quality trials are therefore required to determine whether IPC increases the healing of venous and mixed etiology leg ulcers when used in modern practice where compression therapy is widely used.

Thigh-administered IPC IPC devices usually apply relatively high intermittent pressure over a wound site, which may cause concern to patients and clinicians, may interfere with existing treatments, and may not always be tolerated. A novel IPC device (the WoundExpress, Huntleigh Healthcare) has recently become available on the UK market which could address this issue; the device applies compression to the thigh of the afflicted leg (proximal compression), away from the actual leg ulcer sites which are, by definition, situated below the knee. The device consists of a 3-chamber thigh garment and pneumatic compression pump which delivers a 4-minute compression cycle consisting of a 2-minute venous emptying phase followed by a 2-minute rest phase; it is used for 2 hours per day in a hospital, community or home setting.

A study examined how this thigh IPC device affected distal arterial and venous blood flow in 20 healthy volunteers and 14 patients of leg ulcers of various etiologies. They found that arterial blood flow velocity increased in the dorsalis pedis artery after periods of compression, and that venous blood flow velocity increased when the lower chambers of the cuff deflated; these effects were similar in the healthy volunteers and the patients with leg ulcers. Hence, these results demonstrated that the device resulted in positive effects on venous and arterial blood flow distal to the compression site, but proximal to wound sites.

Further to this, another study conducted a prospective observational pilot study which involved 21 recruited patients with hard to heal wounds utilizing the same thigh administered IPC device for two hours a day for an eight-week period in addition to their standard wound care (hard to heal was defined as failure of the wound to progress in the opinion of the treating clinician and a wound that was observed for an 8 week period prior to recruitment). 95.24% of participants progressed towards healing and pain scores decreased in 83.33%. Most participants felt that the thigh IPC was comfortable and easy to apply and remove in the setting of their own homes. However, this was not a controlled trial with a potential for selection bias.

The IPCOTT study therefore aims to further evaluate the effectiveness of thigh IPC for the treatment of lower limb wounds using gold standard RCT methodology.

Design:

The IPCOTT study is a global, multicenter, pragmatic, open, randomised controlled trial (RCT) of IPC (2hrs daily) plus standard wound care vs. standard wound care alone. One hundred and sixty participants will be recruited across eleven sites which provide wound care in a clinic environment- Aneurin Bevan University Heatlh Board, Cardiff & Vale University Health Board Cwm Taf Morgannwg University Health Board, Wales; Accelerate CIC, London, England; St. Maria Hilf Krankenhaus, Bochum, Germany; Clinique Pasteur, Toulouse, France; Northumbria Healthcare National Health Service Foundation Trust, England; SerenaGroup Monroeville, US), Mid Yorkshire Hospitals National Health Service Trust, England.

Setting:

Eligible patients attending wound clinic appointments at each of the eleven study sites, or patients who have been referred for screening for entry into the study who are found to be eligible, will be invited to participate. Recruitment, consent and all study assessments and data collection will take place in the respective clinics or by a member of the study team visiting the patient in their own home.

Duration of the study: 18 weeks; includes a 2-week run in period followed by 16-week intervention period.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Presence of at least one hard to heal*, venous or mixed (of both venous and arterial origin) aetiology lower limb wound
* ABPI ≥ 0.6, or, where an ABPI measure is not viable, use of locally-approved alternative assessments to rule out significant peripheral arterial disease i.e. doppler auscultation, toe pressure assessment (Absolute Toe Pressure ≥40mmHg ) or arterial imaging
* Has received high static compression therapy (in the form of bandages, wraps or hosiery) during the preceding 4 weeks and is willing to continue receiving appropriate static compression therapy for their ulcer aetiology for the duration of the study
* Receiving standard wound care as per investigator discretion which will continue regardless of study participation
* Able and willing to give informed consent for participation in study
* Able to self-apply IPC garment (supplied) and connect to an electrically operated pump at home for two hours daily for a 16 week period
* Females of childbearing potential must be willing to use acceptable methods of contraception (birth control pills, barriers or abstinence) during the course of the study and undergo a pregnancy test at screening

  * Failure of wound to progress towards healing (as indicated by decrease in surface area by ≥ 25%) in preceding month, despite appropriate and adequate compression therapy.

Exclusion Criteria:

* Wound surface area ≥ 100cm2
* Wound duration ≤ 2 months or ≥ 5 years
* Diabetic patients with recent HbA1c >8.5
* Known or suspected deep vein thrombosis (DVT), pulmonary embolism, thrombophlebitis and acute infections of the skin, such as cellulitis
* Decompensated/severe congestive cardiac failure, pulmonary oedema associated with significant limb oedema or any condition where an increase of fluid to the heart may be detrimental
* Severe arteriosclerosis or other ischemic vascular disease
* Leg ulcers without a venous component to their aetiology (e.g., arterial or rheumatoid) or significant peripheral vascular disease which contraindicates compression (ABI < 0.6 or Absolute Toe Pressure <40mmHg)
* Known malignancy
* Patient receiving any other adjunctive wound therapy such as heat, topical negative therapy, biotherapy
* Current participation in any other clinical trial
* Patient likely to miss more than five days of therapy (e.g. for planned holiday)
* Thigh circumference >90cm (maximum garment size)
* Any wounds, infection or dermatological conditions that would be adversely affected by placement of the thigh garment
* Subject is pregnant or breast-feeding

Ɨ within preceding 3 months

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2023-01-25 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
Determine the effect of thigh administered IPC on the healing of lower limb wounds of venous or mixed etiology | 16 weeks
  Assess percentage change to wound surface area of the reference ulcer following a 16-week intervention period as assessed by the percentage of change in wound surface. This will be calculated using the measurements from wound photographs and by dividing the change by the baseline area. A percentage below zero will indicate an increase in wound size and a percentage above zero indicates a reduction in wound size at week 16 compared with baseline.

SECONDARY OUTCOMES:
Assess the effect of IPC on patient experience of wound related pain | 16 weeks
  Change in patient reported wound related pain as assessed by visual analogue score
Assess the effect of IPC on patient quality of life | 16 weeks
  Change in patient reported quality of life score as assessed by the Cardiff Wound Impact Schedule
Assess patient acceptability of IPC therapy | 16 weeks
  Assess duration of IPC device usage by comparing patient-reported IPC device usage as reported in the patient diary and actual IPC device usage according to the device data logger
Assess the cost effectiveness of IPC as a treatment for venous and mixed etiology leg ulcers | 16 weeks
  EQ5D-5L will be used to derive a patient reported outcome measure for use in the cost-effectiveness analysis.
Determine the proportion of patients with wound closure at week 16 | 16 weeks
  Assess proportion of patients with complete wound healing, defined as complete, full, 100% re-epithelialization or closure without discharge, drainage/scab. Assessed by two blinded assessors from wound photographs and measurements
Assess safety of IPC therapy | 16 weeks
  Assess Device-related adverse events/serious adverse events.

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Royal Research, Hollywood, Florida
  - Three Rivers Wound and Hyperberic, North Port, Florida
  - Wound Care of Tulsa, Tulsa, Oklahoma
  - SerenaGroup, Monroeville, Pennsylvania
  - SerenaGroup Research, Austin, Texas

IPD SHARING:
Plan to Share IPD: Yes
There is a plan to share Individual participant data (IPD). Study protocol, Statistical Analysis Plan (SAP), Informed Consent Form (ICF) Clinical Study Report (CSR) will be shared immediately following publication with open access at www.huntleigh-healthcare.us
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Immediately following publication. No end date.
Access Criteria: Anyone who wishes to access the data
URL: http://huntleigh-healthcare.us

REFERENCES:
- [Background] Aboyans V, Criqui MH, Abraham P, Allison MA, Creager MA, Diehm C, Fowkes FG, Hiatt WR, Jonsson B, Lacroix P, Marin B, McDermott MM, Norgren L, Pande RL, Preux PM, Stoffers HE, Treat-Jacobson D; American Heart Association Council on Peripheral Vascular Disease; Council on Epidemiology and Prevention; Council on Clinical Cardiology; Council on Cardiovascular Nursing; Council on Cardiovascular Radiology and Intervention, and Council on Cardiovascular Surgery and Anesthesia. Measurement and interpretation of the ankle-brachial index: a scientific statement from the American Heart Association. Circulation. 2012 Dec 11;126(24):2890-909. doi: 10.1161/CIR.0b013e318276fbcb. Epub 2012 Nov 16. No abstract available. PMID 23159553
- [Background] Alvarez OM, Wendelken ME, Markowitz L, Comfort C. Effect of High-pressure, Intermittent Pneumatic Compression for the Treatment of Peripheral Arterial Disease and Critical Limb Ischemia in Patients Without a Surgical Option. Wounds. 2015 Nov;27(11):293-301. PMID 26574751
- [Background] Arthur J, Lewis P. When is reduced-compression bandaging safe and effective? J Wound Care. 2000 Nov;9(10):469-71. doi: 10.12968/jowc.2000.9.10.26301. PMID 11933451
- [Background] Arvesen K, Nielsen CB, Fogh K. Accelerated wound healing with combined NPWT and IPC: a case series. Br J Community Nurs. 2017 Mar;22 Suppl 3(Sup3):S41-S45. doi: 10.12968/bjcn.2017.22.Sup3.S41. PMID 28252337
- [Background] Burnand KG, Whimster I, Naidoo A, Browse NL. Pericapillary fibrin in the ulcer-bearing skin of the leg: the cause of lipodermatosclerosis and venous ulceration. Br Med J (Clin Res Ed). 1982 Oct 16;285(6348):1071-2. doi: 10.1136/bmj.285.6348.1071. PMID 6812751
- [Background] Chen AH, Frangos SG, Kilaru S, Sumpio BE. Intermittent pneumatic compression devices -- physiological mechanisms of action. Eur J Vasc Endovasc Surg. 2001 May;21(5):383-92. doi: 10.1053/ejvs.2001.1348. PMID 11352511
- [Background] Comerota AJ. Intermittent pneumatic compression: physiologic and clinical basis to improve management of venous leg ulcers. J Vasc Surg. 2011 Apr;53(4):1121-9. doi: 10.1016/j.jvs.2010.08.059. Epub 2010 Nov 3. PMID 21050701
- [Background] Delis KT, Husmann MJ, Cheshire NJ, Nicolaides AN. Effects of intermittent pneumatic compression of the calf and thigh on arterial calf inflow: a study of normals, claudicants, and grafted arteriopaths. Surgery. 2001 Feb;129(2):188-95. doi: 10.1067/msy.2001.110023. PMID 11174701
- [Background] Dolibog P, Franek A, Taradaj J, Dolibog P, Blaszczak E, Polak A, Brzezinska-Wcislo L, Hrycek A, Urbanek T, Ziaja J, Kolanko M. A comparative clinical study on five types of compression therapy in patients with venous leg ulcers. Int J Med Sci. 2013 Dec 14;11(1):34-43. doi: 10.7150/ijms.7548. eCollection 2014. PMID 24396284
- [Background] Geerts WH, Bergqvist D, Pineo GF, Heit JA, Samama CM, Lassen MR, Colwell CW. Prevention of venous thromboembolism: American College of Chest Physicians Evidence-Based Clinical Practice Guidelines (8th Edition). Chest. 2008 Jun;133(6 Suppl):381S-453S. doi: 10.1378/chest.08-0656. PMID 18574271
- [Background] Giddings, J., Ralis, H., Jennings, G., & McLeod, A. (2001). Suppression of the tissue factor pathway combined with enhanced tissue plasminogen activator activity (tPA) after intermittent pneumatic compression. Journal of Thrombosis and Haemostasis (Supplement), 86, 2240.
- [Background] Guest JF, Ayoub N, McIlwraith T, Uchegbu I, Gerrish A, Weidlich D, Vowden K, Vowden P. Health economic burden that wounds impose on the National Health Service in the UK. BMJ Open. 2015 Dec 7;5(12):e009283. doi: 10.1136/bmjopen-2015-009283. PMID 26644123
- [Background] Guest JF, Ayoub N, McIlwraith T, Uchegbu I, Gerrish A, Weidlich D, Vowden K, Vowden P. Health economic burden that different wound types impose on the UK's National Health Service. Int Wound J. 2017 Apr;14(2):322-330. doi: 10.1111/iwj.12603. Epub 2016 May 26. PMID 27229943
- [Background] Guest JF, Fuller GW, Vowden P. Venous leg ulcer management in clinical practice in the UK: costs and outcomes. Int Wound J. 2018 Feb;15(1):29-37. doi: 10.1111/iwj.12814. Epub 2017 Dec 15. PMID 29243398
- [Background] Husmann M, Willenberg T, Keo HH, Spring S, Kalodiki E, Delis KT. Integrity of venoarteriolar reflex determines level of microvascular skin flow enhancement with intermittent pneumatic compression. J Vasc Surg. 2008 Dec;48(6):1509-13. doi: 10.1016/j.jvs.2008.07.016. Epub 2008 Oct 1. PMID 18829220
- [Background] Kakkos SK, Caprini JA, Geroulakos G, Nicolaides AN, Stansby GP, Reddy DJ. Combined intermittent pneumatic leg compression and pharmacological prophylaxis for prevention of venous thromboembolism in high-risk patients. Cochrane Database Syst Rev. 2008 Oct 8;(4):CD005258. doi: 10.1002/14651858.CD005258.pub2. PMID 18843686
- [Background] Kumar S, Samraj K, Nirujogi V, Budnik J, Walker MA. Intermittent pneumatic compression as an adjuvant therapy in venous ulcer disease. J Tissue Viability. 2002 Apr;12(2):42-4, 46, 48 passim. doi: 10.1016/s0965-206x(02)80013-4. PMID 12001325
- [Background] Lim SLX, Chung RE, Holloway S, Harding KG. Modified compression therapy in mixed arterial-venous leg ulcers: An integrative review. Int Wound J. 2021 Dec;18(6):822-842. doi: 10.1111/iwj.13585. Epub 2021 Mar 18. PMID 33738975
- [Background] McCulloch JM, Marler KC, Neal MB, Phifer TJ. Intermittent pneumatic compression improves venous ulcer healing. Adv Wound Care. 1994 Jul;7(4):22-4, 26. PMID 7827744
- [Background] Mills JL Sr, Conte MS, Armstrong DG, Pomposelli FB, Schanzer A, Sidawy AN, Andros G; Society for Vascular Surgery Lower Extremity Guidelines Committee. The Society for Vascular Surgery Lower Extremity Threatened Limb Classification System: risk stratification based on wound, ischemia, and foot infection (WIfI). J Vasc Surg. 2014 Jan;59(1):220-34.e1-2. doi: 10.1016/j.jvs.2013.08.003. Epub 2013 Oct 12. PMID 24126108
- [Background] Moran PS, Teljeur C, Harrington P, Ryan M. A systematic review of intermittent pneumatic compression for critical limb ischaemia. Vasc Med. 2015 Feb;20(1):41-50. doi: 10.1177/1358863X14552096. Epub 2014 Sep 30. PMID 25270409
- [Background] Morris RJ, Ridgway BS, Woodcock JP. The use of intermittent pneumatic compression of the thigh to affect arterial and venous blood flow proximal to a chronic wound site. Int Wound J. 2020 Oct;17(5):1483-1489. doi: 10.1111/iwj.13418. Epub 2020 Jun 17. PMID 32558254
- [Background] Naik G, Ivins NM, Harding KG. A prospective pilot study of thigh-administered intermittent pneumatic compression in the management of hard-to-heal lower limb venous and mixed aetiology ulcers. Int Wound J. 2019 Aug;16(4):940-945. doi: 10.1111/iwj.13125. Epub 2019 Apr 23. PMID 31016851
- [Background] Nelson EA, Hillman A, Thomas K. Intermittent pneumatic compression for treating venous leg ulcers. Cochrane Database Syst Rev. 2014 May 12;2014(5):CD001899. doi: 10.1002/14651858.CD001899.pub4. PMID 24820100
- [Background] National Clinical Guideline Centre (UK). Varicose Veins in the Legs: The Diagnosis and Management of Varicose Veins. London: National Institute for Health and Care Excellence (NICE); 2013 Jul. Available from http://www.ncbi.nlm.nih.gov/books/NBK264166/ PMID 25535637
- [Background] Persoon A, Heinen MM, van der Vleuten CJ, de Rooij MJ, van de Kerkhof PC, van Achterberg T. Leg ulcers: a review of their impact on daily life. J Clin Nurs. 2004 Mar;13(3):341-54. doi: 10.1046/j.1365-2702.2003.00859.x. PMID 15009337
- [Background] Phillips CJ, Humphreys I, Thayer D, Elmessary M, Collins H, Roberts C, Naik G, Harding K. Cost of managing patients with venous leg ulcers. Int Wound J. 2020 Aug;17(4):1074-1082. doi: 10.1111/iwj.13366. Epub 2020 May 7. PMID 32383324
- [Background] Sayegh, A. (1987). Intermittent pneumatic compression: past, present and future. Clinical Rehabilitation, 1(1), 59-64.
- [Background] Scottish Intercollegiate Guidelines Network. (2010). Management of chronic venous leg ulcers. A national clinical guideline.
- [Background] Schuler JJ, Maibenco T, Megerman J, Ware M, Montalvo J (1996) Treatment of chronic venous ulcers using sequential intermittent pneumatic compression. Phlebology; 11(3): 111-6.
- [Background] Stevens J. Diagnosis, assessment and management of mixed aetiology ulcers using reduced compression. J Wound Care. 2004 Sep;13(8):339-43. doi: 10.12968/jowc.2004.13.8.26661. PMID 15469220
- [Background] Tessari M, Tisato V, Rimondi E, Zamboni P, Malagoni AM. Effects of intermittent pneumatic compression treatment on clinical outcomes and biochemical markers in patients at low mobility with lower limb edema. J Vasc Surg Venous Lymphat Disord. 2018 Jul;6(4):500-510. doi: 10.1016/j.jvsv.2018.01.019. PMID 29909855
- [Background] van Bemmelen PS, Gitlitz DB, Faruqi RM, Weiss-Olmanni J, Brunetti VA, Giron F, Ricotta JJ. Limb salvage using high-pressure intermittent compression arterial assist device in cases unsuitable for surgical revascularization. Arch Surg. 2001 Nov;136(11):1280-5; discussion 1286. doi: 10.1001/archsurg.136.11.1280. PMID 11695973
- [Background] WUWHS (2008) Principles of best practice: compression in venous leg ulcers. A consensus document.
- [Background] Smith PC, Sarin S, Hasty J, Scurr JH. Sequential gradient pneumatic compression enhances venous ulcer healing: a randomized trial. Surgery. 1990 Nov;108(5):871-5. PMID 2237768
- [Result] Mosti G, Iabichella ML, Partsch H. Compression therapy in mixed ulcers increases venous output and arterial perfusion. J Vasc Surg. 2012 Jan;55(1):122-8. doi: 10.1016/j.jvs.2011.07.071. Epub 2011 Sep 23. PMID 21944912